CLINICAL TRIAL: NCT02739854
Title: The Prevalence and Risk Factors for Lung Atelectasis in Patients With Critical Trauma Who Are Intubated and Mechanically Ventilated
Brief Title: Prevalence of Atelectasis in Critical Trauma Patients
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Guntaragorn Hongrattana, Principal Investigator, Khon Kaen University
Other Study IDs: VHI-prevalence-atelectasis
Record Dates: First submitted 2016-01-28; First posted 2016-04-15 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Atelectasis
Keywords: trauma; atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify the prevalence rate and risk factors for pulmonary complications in patients with critical trauma who intubated and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* An inclusion criterion is the traumatic patients (e.g. head injury, blunt chest, blunt abdomen, and fracture of spine; with or without operative, pure or multitrauma) with intubation and mechanical ventilation who admit at this time period will recruit to the study.

Exclusion Criteria:

* a patients who admit less than 1 day will be excluded such as sudden death or moving to other ward because of improving conditions, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The critically traumatic patients who were admitted to the traumatic surgical intensive care unit at Khon Kaen Hospital (February 2016 to February 2017).
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
number of participants with pulmonary atelectasis | from the date of randomization until the date of first documented of atelectasis, assessed up to 1 years

SECONDARY OUTCOMES:
number of participants with pneumonia | from the date of randomization until the date of first documented of pneumonia, assessed up to 1 years
number of participants with pleural effusion | from the date of randomization until the date of first documented of pleural effusion, assessed up to 1 years
number of participants with abnormal laboratory values | from the date of randomization until the date of first documented of pleural effusion, assessed up to 1 years
  the laboratory test include arterial blood gases (ABG), Clinical chemistry test (i.e. Blood urea nitrogen, Creatinine, Sodium, Potassium, Phosphorus, Chloride, Magnesium).
number of participants with adverse events that are related to treatment | from the date of randomization until the date of first documented of pleural effusion, assessed up to 1 years
  These data are collected from medical records (i.e. arrhythmia, hypoxia)

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand